CLINICAL TRIAL: NCT05573191
Title: Effects of Intravenous Lidocaine on ED50, ED95 and NTI Values of Propofol Induced Unconsciousness
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Principal Investigator, Hanxiang Ma, Director of department, General Hospital of Ningxia Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: JGM 20220123
Record Dates: First submitted 2022-09-30; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: General Anesthesia
Keywords: ED50; ED95; intravinious lidocaine; propofol; NTI
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LP group (Experimental): The experimental group received 1.5 mg/kg lidocaine intravenously,after 90s, the corresponding dose of propofol was injected intravenously at 30mg/kg/h, and to observe Whether consciousness disappears or not，recording NTI values, heart rate, oxygen saturation, mean arterial pressure and drug side effects in the baseline state, 90s after lidocaine administration, 60s and 120s after propofol administration
  Interventions: Drug: Lidocaine
- P group (Placebo Comparator): Replace lidocaine with equal volume normal saline,Others are the same as the experimental group.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — The experimental group was injected with lidocaine 1.5mg/kg, and propofol was pumped intravenously at 90s after lidocaine injection.The dose of propofol was further set according to groups. The heart rate, mean arterial pressure, pulse oxygen saturation and NTI values of subjects were recorded in tne basic state,during the 90s after lidocaine administration, 60s after propofol administration and consciousness loss.The control group simply replaced lidocaine with equal volume normal saline
  Arms: LP group
Drug: Normal saline — Normal saline
  Arms: P group

SUMMARY:
The effect of intravenous lidocaine on ED50 and ED95 of propofol, which causes unconsciousness, is unclear. In addition, it is not clear whether the depth of anesthesia induced by propofol changes when lidocaine is used in combination. Therefore, the purpose of this study was to study the effects of intravenous lidocaine on ED50, ED95 and NTI values of propofol induced unconsciousness .

DETAILED DESCRIPTION:
Intravenous lidocaine has many advantages in perioperative period, in addition to reducing the amount of opioids and propofol, thus reducing the incidence of adverse reactions caused by them, it also has the effect on organ protection, can shorten the length of hospital stay, and promote postoperative recovery. The effect of intravenous lidocaine on ED50 and ED95 of propofol, which causes unconsciousness, is unclear. In addition, it is not clear whether the depth of anesthesia induced by propofol changes when lidocaine is used in combination. Therefore, the purpose of this study was to study the effects of intravenous lidocaine on ED50, ED95 and NTI values of propofol induced unconsciousness .

ELIGIBILITY:
Inclusion Criteria:

1. The informed consent is signed
2. Aged 18 to 65 years old
3. ASA is rated from I to II
4. Body mass index ranged from 18.5 to 24.9 kg/m2

Exclusion Criteria:

1. Unwilling to sign informed consent or refuse to participate in the study
2. Patients with serious arrhythmia and organic heart disease before surgery
3. Sedative and analgesic drugs were taken within 1 week before surgery
4. Lidocaine allergy
5. Patients with mental and neurological diseases
6. Patients with difficult airway
7. People with hearing impairment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-08 (Estimated); Primary Completion 2022-11-08 (Estimated); Study Completion 2022-11-25 (Estimated)

PRIMARY OUTCOMES:
The number of patients with loss of consciousness | 6 hours
  Effects of intravenous lidocaine on ED50 and ED95 of propofol induced unconsciousness

SECONDARY OUTCOMES:
Effects of intravenous lidocaine on NTI values of propofol induced unconsciousness | 6 hours
  The NTI values at T1,T2,T3 and T4 were recorded and statistically analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Guimei Ji, master, Principal Investigator — General Hospital of Ningxia Medical University
Locations (2):
- China (2):
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - GuiMei Ji, Yinchuan, Ningxia